CLINICAL TRIAL: NCT01492985
Title: Evaluation of a Therapeutic Immunization Strategy Associating a DNA Vaccine (GTU-MultiHIV B) Followed by a Lipopeptide Vaccine (LIPO-5) in the Control of Viral Replication Following Antiretroviral Treatment Interruption in HIV-1 Infected Patients With a CD4 Cell Count ≥ 600/mm3
Brief Title: Lipopeptide Immunisation With GTU-multiHIV Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-018198-30; ANRS 149 LIGHT (Other: ANRS)
Record Dates: First submitted 2011-11-24; First posted 2011-12-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-02

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine placebos (Placebo Comparator): Vaccine placebos corresponding to the dilutant of these vaccines
  Interventions: Biological: Placebos of GTU-multiHIV B and LIPO-5 vaccines
- Vaccine arm (Experimental)
  Interventions: Biological: GTU-multHIV B vaccine and LIPO-5 vaccine

INTERVENTIONS:
Biological: Placebos of GTU-multiHIV B and LIPO-5 vaccines — Placebos corresponds respectively to 1X PBS pH = 7.2 and glucose 5%
  Arms: Vaccine placebos
Biological: GTU-multHIV B vaccine and LIPO-5 vaccine — Vaccines are respectively an HIV-DNA plasmid and a mixture of 5 HIV-lipopeptides.
  Arms: Vaccine arm

SUMMARY:
The combination of GTU-MultiHIV B DNA and LIPO-5 vaccines in a prime-boost strategy is expected to induce strong and diverse HIV-specific immune responses in HIV-infected patients. The investigators will carry out the clinical therapeutic immunization "proof of concept" trial in HIV infected patients. The investigators propose a multi-center double blind randomized versus placebo phase II clinical trial in patients who are chronic asymptomatic HIV-infected patients, with undetectable viral load while treated with a potent combination of antiviral drugs. Patients will continue antiviral therapy combined with either therapeutic vaccination or placebo vaccination. Patients will undergo the procedure which includes a prime with the GTU-MultiHIV B DNA vaccine or placebo administered by IM injections via Biojector (a needle-free injection system) followed by a boost of LIPO-5 vaccine or placebo also given IM.

In total, 105 HIV-1 patients will be enrolled: 35 in the placebo arm and 70 in the vaccine arm. Patients will receive antiretroviral treatments and 3 administrations of DNA vaccine or its placebo at weeks 0, 4 and 12 (corresponding to prime vaccinations). They also receive 2 doses of LIPO-5 vaccines or its placebo at week 20 and 24 (corresponding to boost vaccinations). At week 36 antiretroviral treatments will be interrupted until week 48. Patients will be intensely monitored during the treatment interruption period. After start of cART treatment (at the latest in W48), a data collection from clinical car will be carried out. A blood sample with W74 will allow to study the persistence ot the immunizing responses, 1 year after the injection of the last vaccine/placebo.

The primary efficacy endpoint is a plasma HIV-1 RNA level at week 48 (e.g. 12 weeks after stopping all antiviral treatment).

The main hypothesis for conducting a phase II randomized trial is that immune responses in vaccinated patients may be associated with a better control of viral replication following c-ART interruption as compared to placebo-vaccinated patients.

ELIGIBILITY:
Inclusion criteria:

* Documented HIV-1 infection (ELISA and Western blot)
* Age ≥ 18 years and < 60 years
* No history of CDC category C clinical events (1993), including cutaneous Kaposi's sarcoma
* CD4 Nadir ≥ 300/mm3 Under antiretroviral treatment
* CD4 ≥ 600/mm3 on all measurements within the previous 6 months* prior to W-3 screening visit (one single CD4 value between 550-600 cells/ mm3 is permitted)
* CD4 value ≥ 600/ mm3 at W-3 screening visit
* Plasma HIV1-RNA < 50 copies/mL on all measurements within the previous 6 months* (An occasional measurement of HIV-1 RNA (so-called " blip " between 50 and 200 copies/mL is permitted)
* HIV1-RNA < 50 copies/mL at W-3 screening visit

  * In the absence of measurement in the last 6 months, a measurement performed in the last 12 months is accepted
* Treatment with a combination of antiviral drugs (cART) for at least 18 months regardless of the combination, under condition that :

  * in the W24 visit the non-nucleoside inhibitors are replaced by a protease inhibitor potentiated by ritonavir
  * no failure or resistance to the protease inhibitor was previously reported
* With adequate method of contraception and negative pregnancy test (βHCG plasma) for women of childbearing potential
* Laboratory parameters at W-3:

  * polynuclear neutrophils ≥ 1,000/mm3
  * haemoglobin ≥ 10 g/dl
  * platelets ≥ 100,000/mm3
  * creatinine ≤ 1.5 x N
  * AST, ALT, bilirubin ≤ 2.5 x N
  * proteinuria ≤ 1 g/L (++)
  * anti-nuclear antibodies ≤ 1/320
  * anticardiolipin antibodies ≤ 30 U
  * no lupus anticoagulant
* Participant agreeing to be treated and followed for at least 74 weeks according to the protocol
* Participant agreeing to interrupt his/her cART treatment and, if applicable, to replace the non-nucleoside inhibitors by a protease inhibitor potentiated by ritonavir at W24
* Participant agreeing to the use of condom, in particular during ART interruption period (between the visit S36 and the visite S48)
* Participant covered by HealthInsurance (article L1121-11 of Code de la Santé Publique)
* Written informed consent (at the latest the day of pre-inclusion and before all exams to be done in the context of the trial) (article L1122-1-1 of Code de la Santé Publique).

Exclusion criteria

* Pregnancy or lactation,
* HIV-2 infection (isolated or associated with HIV-1),
* History of (experimental) vaccinations against HIV,
* Treatment with chemotherapy or interferon alpha (IFN-α-2b), sargramostim (GM-CSF), IL-2 or IL-7 ongoing or in the previous12 weeks before inclusion (W0),
* Treatment with corticoids or immunosuppressive agents ongoing or in the previous12 weeks before inclusion in the trial (W0),
* Administration of a live vaccine within 60 days prior to inclusion in the trial (W0) or any other inactivated vaccine within 14 days before W0 visit
* Planned administration, during the follow-up of participants, of a vaccine other than those recommended in France as part of the usual care of patients
* History of cancer (except basal cellular skin carcinoma),
* History of cardiovascular disease (angina, myocardial infarction, transient ischemic attack, stroke),
* History of renal failure related to HIV,
* History of thrombocytopenia related to HIV (<50,000/mm3),
* Ongoing cardiac, pulmonary, thyroid, renal or neurological (peripheral or central) diseases,
* Progressive infection,
* Co-infection with hepatitis B (HBsAg + or isolated anti-HBc antibodies +) or hepatitis C (anti-HCV antibody and PCR +),
* Known allergy to aminoglycosides,
* Person placed under juridical protection (article L1122-2 of Code de la Santé Publique)
* Person participating in another biomedical research with an exclusion period always ongoing at screening.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-04-08 (Actual)

PRIMARY OUTCOMES:
Plasma HIV-1 RNA level | week 48 (W48)

SECONDARY OUTCOMES:
Plasma HIV-RNA after stopping antiviral treatment | W40, W44, W48 and W74
Percentage of patients with plasma HIV-RNA below 10 000 copies/mL | W48
Ultrasensitive proviral DNA | W-3, W20, W32 and W44
CD4 T cell counts | W40, W44 and W48 or prior HAART resumption and W74
Percentages of patients who resumed HAART | between W36 and W48
Percentages of patients who reached CD4 cell counts < 350/mm3 confirmed two weeks apart | between W36 and W48
Strength of HIV-specific CD4/CD8 responses | W0, W16, W28, W48 or at the time of failure anw W74
Proportion of responders to at least one HIV peptide pool | W0, W16, W28, W48 or at the time of failure and W74
Breadth of CD4/CD8+ HIV-specific responses defined as the number of HIV pools recognized among the 18 pools | W0, W16, W28, W48 or at the time of failure and W74
Polyfunctionality of HIV specific T cell responses evaluated by the mean proportion of CD4/CD8+ T cells producing IL-2 and/or IFN-g following ex-vivo stimulation with HIV-1 peptide pools | W0, W16, W28, W48 and W74
Adverse Events > grade 2 | W0, W4, W12, W16, W20, W24, W28, W32, W36, W38, W40, W42, W44, W48 and W74
AIDS-defining events and serious non-AIDS events defined as cardiovascular diseases, kidney diseases, end stage liver diseases, non-AIDS defining malignancies except basal cellular skin cancer, and bacterial infections | W0, W4, W12, W16, W20, W24, W28, W32, W36, W38, W40, W42, W44, W48 and W74
Analysis of predictive factors for plasma HIV-RNA | W48

CONTACTS AND LOCATIONS:
Overall Officials: Yves Lévy, PU-PH, Principal Investigator — Hôpital Henri Mondor - Créteil - France; Geneviève Chêne, PU-PH, Study Director — CMG-EC de l'INSERM U897 / ANRS
Locations (1):
- Service d'Immunologie clinique, Centre de vaccination anti-VIH ANRS Mondor Ile-de-France, Hôpital Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Alexandre M, Prague M, Lhomme E, Lelievre JD, Wittkop L, Richert L, Levy Y, Thiebaut R. Definition of Virological Endpoints Improving the Design of HIV Cure Strategies Using Analytical Antiretroviral Treatment Interruption. Clin Infect Dis. 2024 Dec 17;79(6):1447-1457. doi: 10.1093/cid/ciae235. PMID 38819800
- [Derived] Levy Y, Lacabaratz C, Lhomme E, Wiedemann A, Bauduin C, Fenwick C, Foucat E, Surenaud M, Guillaumat L, Boilet V, Rieux V, Bouchaud O, Girard PM, Molina JM, Morlat P, Hocqueloux L, Richert L, Pantaleo G, Lelievre JD, Thiebaut R. A Randomized Placebo-Controlled Efficacy Study of a Prime Boost Therapeutic Vaccination Strategy in HIV-1-Infected Individuals: VRI02 ANRS 149 LIGHT Phase II Trial. J Virol. 2021 Apr 12;95(9):e02165-20. doi: 10.1128/JVI.02165-20. Print 2021 Apr 12. PMID 33568510